CLINICAL TRIAL: NCT07234435
Title: Examining the Relationship Between Physical Activity, Nutrition Knowledge, and Burnout Levels of Professionals Serving Individuals With Special Needs and Their Quality of Life
Brief Title: Professionals Serving Individuals With Special Needs and Quality of Life
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Nigde Omer Halisdemir University
Other Study IDs: Special Needs and Professional
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Physiotherapist; Teachers
Keywords: Nutrition knowledge level; individuals with special needs; physical activity; burnout; quality of life
MeSH Terms: conditions — Motor Activity; Burnout, Psychological | interventions — Maslach Burnout Inventory

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Professionals Serving Individuals with Special Needs: The difficulty and slow progress of programs implemented for individuals with special needs can cause physical and emotional wear and tear on professionals providing services to individuals, change in their eating habits, decrease their quality of life, and affect their general health.
  * Physiotherapists, occupational therapists, and teachers working in a private education and rehabilitation center or any public institution.
  * Physiotherapists, occupational therapists, and teachers who have been working for at least two years, due to professional experience and allowance for attrition.
  Interventions: Behavioral: International Physical Activity Questionnaire; Behavioral: The Nutrition Knowledge Level Scale; Behavioral: Maslach Burnout Inventory; Behavioral: Short Form-36 Health Survey

INTERVENTIONS:
Behavioral: International Physical Activity Questionnaire — The physical activity levels of the participants will be assessed using the International Physical Activity Questionnaire (IPAQ). In this study, the self-administered short form, which covers the last seven days, will be used.
  The total score of the questionnaire is calculated by summing the duration (in minutes) and frequency (in days) of walking, moderate, and vigorous activities. .
Behavioral: The Nutrition Knowledge Level Scale — It is assumed that nutritional knowledge enables individuals to choose healthy foods, prepare them in accordance with healthy eating recommendations, and consume them appropriately, thereby leading to improvements in dietary habits. The Nutrition Knowledge Level Scale for Adults, recently developed by Batmaz and Güneş (2018) in Turkey, includes subdomains such as basic nutrition and dietary preferences (Batmaz, H., & Güneş, E., 2018).
Behavioral: Maslach Burnout Inventory — Burnout levels will be assessed using the Maslach Burnout Inventory (MBI). Developed by Maslach and Jackson (1981), the inventory conceptualizes burnout not as a single-dimensional construct but as a multifaceted phenomenon, allowing each dimension to be evaluated independently rather than by a single overall score. The MBI consists of 22 items grouped under three subscales: Emotional Exhaustion, Depersonalization, and Personal Accomplishment.
Behavioral: Short Form-36 Health Survey — Quality of life will be assessed using the Short Form-36 Health Survey (SF-36). This is a self-report questionnaire that evaluates eight dimensions of health through 36 items: physical functioning, social functioning, role limitations due to physical and emotional problems, mental health, vitality (energy), bodily pain, and general health perception.

SUMMARY:
In recent years, the number of individuals with special needs (SNIs) requiring care has been increasing both globally and in our country. In line with the principles of a social welfare state, professionals have taken on a growing role in the care, treatment, and education of SNIs. These professionals include physiotherapists, teachers, psychologists, occupational therapists, and social workers. Unlike the education and treatment of typically developing individuals, providing services to SNIs can place additional burdens on staff, potentially leading over time to various physical, psychological, and emotional challenges. The demanding nature of working with SNIs, high expectations, environmental conditions, low wages despite intensive labor, lack of job security in the private sector, and the potential risks associated with working with individuals with disabilities can all create significant stress for service providers. This, in turn, may negatively affect both their personal and family lives as well as the quality of the services delivered.

DETAILED DESCRIPTION:
The demanding nature of working with SNIs, high expectations, environmental conditions, low wages despite intensive labor, lack of job security in the private sector, and the potential risks associated with working with individuals with disabilities can all create significant stress for service providers. This, in turn, may negatively affect both their personal and family lives as well as the quality of the services delivered.

Therefore, this study aims to examine the levels of physical activity, nutritional knowledge, burnout, and quality of life among professionals-such as physiotherapists, special education teachers, and other specialists (e.g., occupational therapists, speech and language therapists)-who provide services to individuals with special needs. Within the scope of the research, physical activity levels will be assessed using the International Physical Activity Questionnaire (IPAQ), nutritional knowledge using the Nutrition Knowledge Questionnaire, burnout levels using the Maslach Burnout Inventory (MBI), and quality of life using the Short Form-36 Health Survey (SF-36). Additionally, informative sessions will be conducted to promote social participation, collaboration, and knowledge exchange among professionals serving individuals with special needs.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Physiotherapists, occupational therapists, and teachers working in a private education and rehabilitation center or any public institution.
* Physiotherapists, occupational therapists, and teachers who have been working for at least two years due to professional experience and attrition.

Exclusion Criteria:

* Individuals who do not volunteer to participate in the study.
* Retired physiotherapists, occupational therapists, and teachers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Professionals who work with individuals with special needs: Physiotherapists, occupational therapists, and teachers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire | 4 months
  The physical activity levels of the participants will be assessed using the International Physical Activity Questionnaire (IPAQ). In this study, the self-administered short form, which covers the last seven days, will be used. The total score of the questionnaire is calculated by summing the duration (in minutes) and frequency (in days) of walking, moderate, and vigorous activities. The time spent sitting (sedentary behavior) is computed separately as an independent score. By multiplying the duration (minutes), frequency (days), and corresponding MET value (metabolic equivalent of task; the ratio of work metabolic rate to resting metabolic rate), a composite score is obtained and expressed as MET-minutes/week. The MET values are defined as 3.3 METs for walking, 4 METs for moderate-intensity activity, and 8 METs for vigorous-intensity activity. Inactive: <600 MET-min/week Low physical activity level: 600-3000 MET-min/week Sufficient physical activity level: >3000 MET-min/week
The Nutrition Knowledge Level Scale | 4 months
  It is assumed that nutritional knowledge enables individuals to choose healthy foods, prepare them in accordance with healthy eating recommendations, and consume them appropriately, thereby leading to improvements in dietary habits. The Nutrition Knowledge Level Scale for Adults, recently developed by Batmaz and Güneş (2018) in Turkey, includes subdomains such as basic nutrition and dietary preferences (Batmaz, H., & Güneş, E., 2018). The scale was developed to assess adults' nutritional knowledge and consists of items addressing food and nutrient knowledge, food preparation and cooking methods, and the relationship between nutrition and health. The items are rated on a five-point Likert scale, ranging from strongly agree (4 points) to strongly disagree (0 points). Items containing incorrect statements regarding nutrition knowledge are reverse scored.
Maslach Burnout Inventory | 4 months
  Burnout levels will be assessed using the Maslach Burnout Inventory (MBI). Developed by Maslach and Jackson (1981), the inventory conceptualizes burnout not as a single-dimensional construct but as a multifaceted phenomenon, allowing each dimension to be evaluated independently rather than by a single overall score. The MBI consists of 22 items grouped under three subscales: Emotional Exhaustion, Depersonalization, and Personal Accomplishment. These subscales collectively assess the degree of burnout experienced by individuals in professional settings. Each item of the Maslach Burnout Inventory (MBI) is rated on a 5-point Likert scale (0 = never, 4 = always). Higher Emotional Exhaustion and Depersonalization scores indicate greater burnout, while higher Personal Accomplishment scores indicate lower burnout. Burnout is evaluated based on the three subscale scores rather than a total score.
Short Form-36 Health Survey | 4 months
  Quality of life will be assessed using the Short Form-36 Health Survey (SF-36). This is a self-report questionnaire that evaluates eight dimensions of health through 36 items: physical functioning, social functioning, role limitations due to physical and emotional problems, mental health, vitality (energy), bodily pain, and general health perception. Each subscale is scored from 0 to 100, with higher scores indicating better perceived health status and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Öztürk, M. (2005). A research on reliability and validity of international physical activity questionnaire and determination of physical activity level in university students. Hacettepe University Health Science Institute an Unpublished PhD Thesis, Ankara (in Turkish).